CLINICAL TRIAL: NCT01212822
Title: Phase II Trial of Pre-operative Bevacizumab and FOLFOX Chemotherapy in Locally Advanced Esophageal Cancer
Brief Title: Bevacizumab and Combination Chemotherapy Before Surgery in Treating Patients With Locally Advanced Esophageal or Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-GI-029; NCI-2013-00603 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB#10-022; FER-GI-029 (Other: Fox Chase Cancer Center); P30CA006927 (NIH)
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Gastroesophageal Junction; Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Squamous Cell Carcinoma of the Esophagus; Stage IA Esophageal Cancer; Stage IA Gastric Cancer; Stage IB Esophageal Cancer; Stage IB Gastric Cancer; Stage IIA Esophageal Cancer; Stage IIA Gastric Cancer; Stage IIB Esophageal Cancer; Stage IIB Gastric Cancer; Stage IIIA Esophageal Cancer; Stage IIIA Gastric Cancer; Stage IIIB Esophageal Cancer; Stage IIIB Gastric Cancer; Stage IIIC Esophageal Cancer; Stage IIIC Gastric Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Stomach Neoplasms | interventions — Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bevacizumab, FOLFOX) (Experimental): NEOADJUVANT THERAPY: Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive FOLFOX chemotherapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46 hours on days 1-2. Treatment with bevacizumab repeats every 2 weeks for 4 courses and treatment with FOLFOX repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  SURGERY: Patients then undergo planned surgical resection 4-6 weeks after 6 courses of chemotherapy and at least 8 weeks since the last dose of bevacizumab.
  ADJUVANT THERAPY: Beginning 8-10 weeks after surgery, patients receive bevacizumab IV, oxaliplatin IV, leucovorin calcium IV, and fluorouracil IV as in neoadjuvant therapy. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Procedure: therapeutic conventional surgery — Undergo surgical resection
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot phase II trial studies how well giving bevacizumab and combination chemotherapy together before surgery works in treating patients with locally advanced esophageal or stomach cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, and oxaliplatin work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab and combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate two-year disease-free survival in patients with resectable esophageal and gastroesophageal (GE) junction cancer treated with perioperative bevacizumab and leucovorin calcium, fluorouracil, and oxaliplatin (FOLFOX).

SECONDARY OBJECTIVES:

I. To assess, by pathological examination after surgical resection, complete and partial response to neoadjuvant therapy.

II. To characterize overall and progression free survival. III. To compare baseline and post-chemotherapy/bevacizumab tissues for biomarkers predicting response or resistance to this approach.

IV. To investigate safety in this setting.

OUTLINE:

NEOADJUVANT THERAPY: Patients receive bevacizumab intravenously (IV) over 30-90 minutes on day 1. Patients also receive FOLFOX chemotherapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46 hours on days 1-2. Treatment with bevacizumab repeats every 2 weeks for 4 courses and treatment with FOLFOX repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

SURGERY: Patients then undergo planned surgical resection 4-6 weeks after 6 courses of chemotherapy and at least 8 weeks since the last dose of bevacizumab.

ADJUVANT THERAPY: Beginning 8-10 weeks after surgery, patients receive bevacizumab IV, oxaliplatin IV, leucovorin calcium IV, and fluorouracil IV as in neoadjuvant therapy. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy proven adenocarcinoma, squamous cell carcinoma or undifferentiated carcinoma of the esophagus, GE junction and/or gastric cardia
* Patients must have potentially resectable disease by the thoracic, minimally invasive or transhiatal approach

  * No portion of the lesion may be within 5 cm of the cricopharyngeus
  * Patient must be considered medically fit for surgery with average or below average risk
  * T1-3 or T4 with local invasion confined to diaphragm, pleura or pericardium
  * No myocardial infarction within 12 months of enrollment
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* White blood cells (WBC) >= 3,500/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine (Cr) =< 1.5 mg and/or creatinine clearance >= 60 cc/min
* Bilirubin must be < upper limit of normal (ULN) unless the patient has a chronic grade 1 bilirubin elevation due to Gilbert's disease or similar syndrome due to slow conjugation of bilirubin
* Alkaline phosphatase must be < ULN
* Aspartate aminotransferase (AST) & alanine aminotransferase (ALT) must be < ULN
* Urine protein/creatinine (UPC) ratio of < 1.0 or dipstick for protein of < 2+, Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v 4) grade < 2; patients with a UPC ratio >= 1.0 or dipstick of 2+ must undergo a 24-hour urine collection and must demonstrate < 1 gm of protein in order to participate
* Patients must give written informed consent and Health Insurance Portability and Accountability Act (HIPAA) consent

Exclusion Criteria:

* Patients with prior chemotherapy for any malignant disorder, thoracic radiotherapy or prior surgical resection of an esophageal tumor are ineligible
* Patients with biopsy-proven invasion of the tracheobronchial tree or tracheo-esophageal fistula are ineligible
* Patients with a history of a curatively treated malignancy must be disease-free for at least two years and have a survival prognosis that is greater than five years
* Eligible patients of reproductive potential (both sexes) must agree to use an accepted and effective method of contraceptive during study therapy and for at least 6 months after the completion of bevacizumab; women must not be pregnant or breast-feeding because the study drugs administered may cause harm to an unborn fetus or breastfeeding child; all females of childbearing potential must have a serum pregnancy test to rule out pregnancy within 7 days prior to registration
* Patients with a history of hypertension must measure < 150/90 mmHg and be on a stable regimen of anti-hypertensive therapy; patients with a history of hypertension who have a blood pressure of 150/90 mmHg, or greater are not eligible; patients with a history of hypertension who have a blood pressure of < 150/90 mmHg but are not on a stable regimen of anti-hypertensive therapy, are not eligible
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Association (NYHA) grade II or greater congestive heart failure
* Patients must not have a serious or non-healing wound, skin ulcers or unhealed bone fracture, or known human immunodeficiency virus (HIV) infection
* Patients with >= grade 2 neuropathy are not eligible
* Patients must not have had significant traumatic injury within 28 days prior to randomization
* Patients with PT (INR) > 1.5 are not eligible; the patient may not be receiving full-dose anticoagulation; prophylactic or full dose anticoagulation are permitted post-resection or for treatment of an intercurrent thrombotic event
* Patients with non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude any of the study therapy drugs are not eligible; specifically excluded are the following conditions: current symptomatic arrhythmia, symptomatic peripheral vascular disease
* Patients with a history of the following within 12 months of study entry are not eligible: arterial thromboembolic events, unstable angina
* Any history of stroke or transient ischemic attack
* Significant vascular disease (i.e. aortic dissection, aortic aneurysm)
* Patients with psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude them from meeting the study requirements are not eligible
* Distant metastases
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Known hypersensitivity to any component of bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04-27 (Actual); Primary Completion 2014-10-24 (Actual); Study Completion 2018-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Denlinger, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Case Western Reserve University, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Bevacizumab, FOLFOX): NEOADJUVANT THERAPY: Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive FOLFOX chemotherapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46 hours on days 1-2. Treatment with bevacizumab repeats every 2 weeks for 4 courses and treatment with FOLFOX repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  SURGERY: Patients then undergo planned surgical resection 4-6 weeks after 6 courses of chemotherapy and at least 8 weeks since the last dose of bevacizumab.
  ADJUVANT THERAPY: Beginning 8-10 weeks after surgery, patients receive bevacizumab IV, oxaliplatin IV, leucovorin calcium IV, and fluorouracil IV as in neoadjuvant therapy. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  bevacizumab: Given IV
  oxaliplatin: Given IV
  leucovorin calcium: Given IV
  fluorouracil: Given IV
  therapeutic conventional surgery: Undergo surgical resection
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Bevacizumab, FOLFOX)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Bevacizumab, FOLFOX)
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  30-39 | 1
  40-49 | 1
  50-59 | 6
  60-69 | 5
  70-79 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: To investigate 2 year disease free survival in pts with resectable esophageal and GE junction cancer treated with perioperative bevaciumab and FOLFOX
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bevacizumab, FOLFOX)
Number analyzed (Participants) | 20
Participants | 4

2. Secondary Outcome: Complete and Partial Response to Neoadjuvant Therapy Based on the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: To assess, by path examination after surgical resection, complete and partial response to neoadjuvant therapy. Characterized using proportions and 95% confidence intervals.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Treatment (Bevacizumab, FOLFOX)
Number analyzed (Participants) | 20
percent of patients | 44.4 [21.5 to 69.2]

3. Secondary Outcome: Overall Survival
Description: Characterized using Kaplan-Meier curves.
Time Frame: 4.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Bevacizumab, FOLFOX)
Number analyzed (Participants) | 20
months | 26.0 [23.7 to 51.4]

4. Secondary Outcome: Progression Free Survival
Description: Characterized using Kaplan-Meier curves. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions and a 5 mm absolute increase, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 3 years
Population: One patient who was not evaluated for progression was excluded from PFS analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Bevacizumab, FOLFOX)
Number analyzed (Participants) | 19
months | 19.0 [13.1 to NA] — insufficient number of participants with events

5. Other Pre Specified Outcome: Change in Biomarker Levels
Description: Means, medians, and standard deviations of the biomarker levels and change in biomarker levels within groups defined by response/resistance outcomes will be reported.
Time Frame: Baseline up to day of surgery
Population: Exploratory endpoint, data is not available for analyses
Arm/Group | Treatment (Bevacizumab, FOLFOX)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed up to 4.5 years. Serious Adverse Events and Other (Not Including Serious) Adverse Events were assessed up to 6 weeks after treatment
Arm/Group | Treatment (Bevacizumab, FOLFOX)
All-Cause Mortality (participants affected / at risk) | 10/20
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bevacizumab, FOLFOX) (N=20)
Nausea (Gastrointestinal disorders) | 3
Vomitting (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Dehydration (General disorders) | 1
Esophageal pain and obstruction (Gastrointestinal disorders) | 1
Low potassium (Investigations) | 1
Pancolitis (Gastrointestinal disorders) | 1
c. difficile infection (Infections and infestations) | 1
Leg numbness and loss of right upper extremity motor strength (Nervous system disorders) | 1
Fever (General disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Purulent drainage (Infections and infestations) | 1
Esophageal fistula (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Loss of appetite (Metabolism and nutrition disorders) | 1
methicillin-susceptible Staphylococcus aureus (Infections and infestations) | 1
Bacteremia (Infections and infestations) | 1
Tri-cupsid endocarditis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bevacizumab, FOLFOX) (N=20)
Anemia (Blood and lymphatic system disorders) | 16
Neutrophil count decreased (Investigations) | 10
Platelet count decreased (Investigations) | 10
White blood cell decreased (Investigations) | 10
Fatigue (General disorders) | 17
Hypoalbuminemia (Metabolism and nutrition disorders) | 17
Nausea (Gastrointestinal disorders) | 10
Neuropathy/paresthesia (Nervous system disorders) | 13
Pain (General disorders) | 13
Diarrhea (Gastrointestinal disorders) | 12
Weight loss (Metabolism and nutrition disorders) | 11
Constipation (Gastrointestinal disorders) | 9
Dysphagia (Gastrointestinal disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 6
Vomitting (Gastrointestinal disorders) | 5
Hypertension (Vascular disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysguesia (Nervous system disorders) | 4
Fever (General disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hyperbilirubinemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Stomasitis (Gastrointestinal disorders) | 3
Depression (Psychiatric disorders) | 2
Edema (General disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Proterinuria (Renal and urinary disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Artery thrombosis (Vascular disorders) | 1
Brachycardia (Cardiac disorders) | 1
Chills (General disorders) | 1
Confusion (Psychiatric disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Eye irritation (Eye disorders) | 1
Hand foot syndrome (Nervous system disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Hemorrhage (General disorders) | 1
Hoarsness (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Substance abuse (Psychiatric disorders) | 1
Thrush (Gastrointestinal disorders) | 1
Alkaline phosphate increased (Investigations) | 4
Aspirate aminotransferase increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 3
Infection without neutropenia (Infections and infestations) | 1
Esophageal dilation (Gastrointestinal disorders) | 1
Esophageal reflux (Gastrointestinal disorders) | 1
Esophageal stenosis (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT01212822/Prot_SAP_000.pdf